CLINICAL TRIAL: NCT07079696
Title: Investigating the Therapeutic Efficacy of All-trans Retinoic Acid in Autism Spectrum Disorder Patients With 15q11-13 Duplication Syndrome
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0465
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-06

CONDITIONS: Dup15q Syndrome; Autism Spectrum Disorder; Therapy; All-trans Retinoic Acid
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group experimental (Experimental): Age: 3-7 years old (stratified into Group 1: 3-5 years; Group 2: 5-7 years).
  Interventions: Drug: ATRA

INTERVENTIONS:
Drug: ATRA — Treatment Phase (Duration: 18 months) Intervention: ATRA oral administration using a stepwise titration protocol (detailed below). Patients may discontinue treatment if intolerable adverse events occur; post-withdrawal symptom exacerbation is monitored.
  *Titration Protocol*
  Treatment Cycle (C): 3 weeks per cycle. Dose escalation follows:
  Cycle Dosage Duration C1.1 15 mg/m²/day 2 weeks on / 1 week off C1.2 20 mg/m²/day 2 weeks on / 1 week off C1.3 25 mg/m²/day 2 weeks on / 1 week off Blinded Assessments: primary endpoints: ADOS-2 SA score, CARS, SRS, ATEC, Gesell, and Sensory Motor (SM) scales.
  Biomarker/Diagnostic tests: blood tests (CBC, liver/kidney function, vitamin panels, ATRA levels, hepatitis markers), neuroimaging (cranial fMRI), neurophysiology (EEG, audiometry), skeletal imaging (limb long-bone radiographs, growth monitoring), and biobanking: 1 blood tube for proteomics (baseline, 6/12/18 months). Repeat all assessments at 6, 12, and 18 months after ATRA treatment.

SUMMARY:
Autism spectrum disorder (ASD) , hereafter referred to as autism, is a group of neurodevelopmental disorders caused by genetic and environmental factors. Its core symptoms are social impairment, repetitive stereotyped behaviors, and restricted interests.

The 15q11-13 region of the human chromosome is a locus prone to structural abnormalities leading to neurological disorders. Maternal duplications within this region lead to Dup15q syndrome , which accounts for approximately 1% of ASD cases .

This region harbors multiple alleles, and current research indicates that the pathophysiological alterations in this syndrome primarily involve UBE3A . Among all genes in the 15q11-13 region, only UBE3A exhibits cell-type-specific maternal monoallelic expression . Consequently, duplication of the UBE3A gene is considered the primary pathogenic factor in the pathology of Dup15q syndrome.

Studies show that the metabolic conversion of retinol to retinoic acid is impaired in ASD patients with UBE3A overexpression and corresponding animal models . Notably, dietary supplementation with all-trans retinoic acid (ATRA) has been shown to significantly ameliorate autism-like behaviors caused by UBE3A overexpression in male mice .

This study aims to evaluate ATRA treatment in children with Dup15q syndrome-related autism , assessing changes in their ADOS-2 scores , to potentially provide a novel therapeutic approach for autism treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical Diagnosis Conducted by two experienced physicians based on Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition （DSM-V）
2. Diagnostic Scale Assessment Performed by professionally certified examiners using ADOS-2
3. Genetic Testing Diagnostic criteria via genomic analysis : detection of 15q11-13 duplication containing UBE3A

Exclusion Criteria:

1. History of acute or chronic infection within the past 3 months
2. Active epileptic seizures within the past 6 months
3. Intake of nutritional supplements (e.g., vitamin A and/or minerals) within the past 1 month
4. History of chronic diseases, including abnormal liver function, abnormal renal function, or thyroid dysfunction

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
ADOS-2 SA score | 6、12、18months after ATRA administration

SECONDARY OUTCOMES:
development scale score | 6、12、18months after ATRA administration

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics, Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, 310009, China., Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided